CLINICAL TRIAL: NCT06543030
Title: Transfemoral Versus Transradial Approach in Transarterial Chemoembolization of Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Adel Abouelmagd Sewisy, M.B.B.CH at Radiology department of Assuit university, Assiut University
Other Study IDs: TACE
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfemoral approach (TFA) group
- Transradial approach (TRA) group

SUMMARY:
Transfemoral Versus Transradial Approach in Transarterial Chemoembolization of Hepatocellular Carcinoma

DETAILED DESCRIPTION:
To compare transfemoral approach (TFA) and transradial approach (TRA) in patients undergoing hepatic chemoembolization in terms of safety, feasibility, and procedural variables, including fluoroscopy time and patient preference.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hepatocellular carcinoma of BCLC (Barcelona Clinic Liver Cancer) stage B
* Also for BCLC stage A patients, in whom ablative therapy has technical limitations.
* Downsizing tumor for resection or transplantation.

Exclusion Criteria:

* Factors related to liver cirrhosis:

  * Decompensated cirrhosis (Child-Pugh B and C, score >8), including jaundice, clinical hepatic encephalopathy, and refractory ascites and/ or hepatorenal syndrome
  * Impaired portal-vein blood flow (portal-vein thrombus, hepatofugal blood flow)
* Factors related to HCC:

  * Extensive tumor involving the entirety of both lobes of the liver
  * Malignant portal vein thrombosis
  * Extra-hepatic metastases
* Impaired renal function:

  * Creatinine ≥2 mg/dl or creatinine clearance <30 ml/min
* Factors related to procedure (Radial artery access):

  * Existing AV (arteriovenous) fistula or graft
  * Pervious major surgery to forearm or wrist
  * Vasculitis
  * Pervious access failure
  * Skin infection or compromised integrity
  * Artery size <2mm
  * Intolerance of hyperextended wrist positioning
  * Severe vasospasm
  * Vessel tortuosity
  * Radial loops
  * Absent or occluded radial artery
  * Atherosclerotic or calcific PAD (peripheral artery disease)
  * Coagulopathy INR>1.5 platelets count <50.000/mmc

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinics of Assuit university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To compare transfemoral approach (TFA) and transradial approach (TRA) in patients undergoing hepatic chemoembolization | Baseline
  To compare transfemoral approach (TFA) and transradial approach (TRA) in patients undergoing hepatic chemoembolization in terms of safety, feasibility, and procedural variables, including fluoroscopy time and patient preference.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospitals, Asyut, Egypt